CLINICAL TRIAL: NCT02006797
Title: Impact of Drug Reconciliation at Discharge and Pharmaceutical Communication Between Hospital and Community Pharmacists on Drug Related Problems: Study Protocol for a Cluster Randomized Cross-over Trial
Brief Title: Communication Between Hospital and Community Pharmacists: Impact on Drug Management at Discharge
Acronym: REPHVIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PREPS12-XP/REPHVIM
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Treatment Error
Keywords: reconciliation; discharge; pharmacist; drug related problems
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): patients with reconciliation procedure at discharge and included in the exchange process
  Interventions: Other: reconciliation
- control (No Intervention): usual care

INTERVENTIONS:
Other: reconciliation — medication reconciliation at discharge and communication of this intervention to patient's community pharmacist
  Arms: intervention

SUMMARY:
This study will evaluate the impact of a communication between hospital pharmacist and community pharmacists in addition to drugs reconciliation procedure at discharge. It will be conducted in 21 french public hospitals.

DETAILED DESCRIPTION:
Transition points during hospitalization are at risk of drug related problems (DRP) especially admission and discharge. Reconciliation procedure at admission lead by a clinical pharmacist had been proved to decrease DRP. The community pharmacist (CP) is often the first health professional that patients meet at discharge. He/she is in charge of dispensing their medication to patients and give treatment information. However because of lack of information community pharmacist is not always able to identify problems and this may lead to dispense wrong drugs and/or wrong dosage and/or give wrong information. The objective of this study is to assess the impact of drug reconciliation performed at discharge completed by a communication between the Hospital Pharmacist (HP) and community pharmacist on drug related problem during the 7 days following discharge at home.

The study is a cluster randomized cross-over trial. It involves 21 French universitarian and non-universitarian hospitals with 42 care units: 22 medical units and 20 surgical units. Each unit (a unit corresponds to a cluster) is involved during two consecutive 14-day periods which are randomly assigned as "experimental" or "control" where control corresponds to usual care. During the experimental period, for each eligible patient discharged during the period, a reconciliation procedure will be performed by the HP, with communication to the patient. The HP will further inform the patient's community pharmacist about patient's drug therapy [modification in home medication, acute drugs prescribed, shelved treatments and/or labs results to survey patient]. Eligible patients will be over 18, attending to the same community pharmacist for at least 3 months. We will exclude patients with a length stay over 21 days (too many therapeutic modifications), those who do not return to home, and also palliative patient. The primary outcome is a composite outcome associating any kind of drug misuse during the 7 days following discharge. It will be assessed by phone at day 7 (+/-2) by a pharmacist in charge of the study (PCS) will phone both patients and community pharmacists . The secondary outcome will be the unplanned hospitalizations observed in each group assessed by phone at day 35 (+/-5). We plan to recruit 1,176 patients, i.e. 14 per period per unit.

This study will assess the impact of a reconciliation procedure at discharge followed by a communication between HP and community pharmacists . Also it will identify the type of patients for which the intervention is the most relevant in France and may be generalized to other countries that have the same care organisation.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18
* patients attending to the same CP for at least 3 months
* patients speaking french

Exclusion Criteria:

* patients with a length stay over 21 days (too many therapeutic modifications),
* patients who do not return to home,
* palliative patients and/or expected end of life
* patients that will not give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1176 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
drug related problems (DRP) | 7 days after patient discharge
  The primary outcome is a composite endpoint associated all the problems/dysfunctions that can be observed from the hospital to home during 7 days after discharge. We will be taking in account the occurence of a dysfunction every time that one of the following problems will happen: - first drug problem; the drug taken by the patient has a problem: it is not the right medicine (Name, form, route, dose). The fault may be 1) an error between the processing of transcription at the admission and the discharge, 2) a therapeutic modification related to therapeutic formulary restriction, the home medication is replaced by an another one that may be less adaptated to patient, 3) an error linked to the writing. Second : patient due to patient; the patient doesn't take what was prescribed and / or treatments that he takes are stopped. Third- :presence of a gap in the continuity and duration of therapy: the patient could not have his medication when he's coming at the pharmacy

SECONDARY OUTCOMES:
all compounds of the composite primary outcome measure (patient errors, medical error and DRP) | day 7 after discharge
clinical impact of problems | days 7 after discharge
  all problems will be scored of the potential iatrogenic impact (from 0: none to 3: fatal) by a team associated a nephrologist, a cardiologist, a gastroenterologist and a clinical pharmacist.
number of non-planned hospitalization | days 35 after discharge
  number of non-planned hospitalizations in each group
patient satisfaction | day 7 after patient discharge
  the patient will have to tell his satisfaction about his drugs management by health professionals at discharge. It will be evaluated by a Likert scale with 4 items.
community pharmacist satisfaction about exchanges with hospital pharmacists | 7 days after patient discharge
  the community pharmacist will have to tell his satisfaction about his drugs management by health professionals at discharge. It will be evaluated by a Likert scale with 4 items.
time spend by hospital pharmacist on reconciliation and communication to community pharmacist | at day 2/3 after discharge
  the hospital pharmacist will notice the time spent to patient reconciliation and communicate informations to community pharmacist. Time will be those declared by the hospital pharmacist
percentage of drugs prescription modified by the hospital pharmacist at discharge | at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Xavier POURRAT, Pr, Study Director — Centre Hospitalier Régional Universitaire de Tours
Locations (21):
- France (21):
  - Centre Hospitalier Alès-Cévennes, Alès
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier, Béthune
  - Centre Hospitalier, Blois
  - Hopital de la Cavale Blanche, Brest
  - Hopital ESTAING, Clermont-Ferrand
  - Hopitaux civils de Colmar, Colmar
  - Centre Hospitalier Compiègne-Noyon, Compiègne
  - Centre Hospitalier Universitaire, Grenoble
  - Hopital Jacques Monod, Le Havre
  - Centre Hospitalier, Le Mans
  - CHU Conception, Marseille
  - Hopital de Mercy Metz-Thionville, Metz
  - Centre Hospitalier Pierre Bérégovoy, Nevers
  - Hopital Archet, Nice
  - Centre Hospitalier, Nîmes
  - Centre Hospitalier Universitaire, Poitiers
  - Hopital Inter Armées, Saint-Mandé
  - Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire, Toulouse
  - Centre Hospitalier Universitaire, Tours

REFERENCES:
- [Derived] Pourrat X, Roux C, Bouzige B, Garnier V, Develay A, Allenet B, Fraysse M, Halimi JM, Grassin J, Giraudeau B. Impact of drug reconciliation at discharge and communication between hospital and community pharmacists on drug-related problems: study protocol for a randomized controlled trial. Trials. 2014 Jun 30;15:260. doi: 10.1186/1745-6215-15-260. PMID 24981605